CLINICAL TRIAL: NCT03305796
Title: Detection of Cholesteatoma Using Diffusion Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amer Ragab Ahmed, Principle Investigator, Assiut University
Other Study IDs: Cholesteatoma
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Cholesteatoma
MeSH Terms: conditions — Cholesteatoma | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Diffusion magnetic resonance imaging — Patients with suspected cholesteatoma will have diffusion magnetic resonance imaging

SUMMARY:
Cholesteatoma is a retraction pocket lined with squamous epithelium lined with keratin debris occurring within pneumatized spaces of the temporal bone. Cholesteatomas have a propensity for growth, bone destruction, and chronic infection.High-resolution computerized tomography is the method of choice for imaging the middle ear .

DETAILED DESCRIPTION:
In patients with recurrent cholesteatoma, computerized tomography can show the extent of cholesteatoma in relation to the ossicles and mastoid process,but computerized tomography has a high negative predictive value if neither a soft-tissue mass nor bony destructions are shown.However, if a soft-tissue mass in the middle ear is seen on computerized tomography, diagnosis of the mass is not possible because cholesteatoma, mucoid secretion, granulation tissue and cholesterol granuloma can not be differentiated from one another on computerized tomography.

Standard magnetic resonance imaging shows tissues better than computerized tomography,Therefore in patients with cholesteatoma, magnetic resonance imaging plays a complementary role to computerized tomography in the diagnostic workup, Although computerized tomography provides excellent Bony resolution for showing the anatomy, magnetic resonance imaging provides specificity in characterizing soft-tissue abnormalities shown on computerized tomography,How ever standard magnetic resonance imaging frequently fails to allow differentiation of cholesteatoma from other soft tissues or mucoid secretions, particularly in patients who had ear surgery.

Recent studies of diffusion weighted magnetic resonance imaging show that it is sensitive to cholesteatoma tissue.Recent studies highlights the ability of diffusion weighted magnetic resonance imaging in differentiating cholesteatoma from granulation tissue in patients who have undergone mastoidectomy and also these imaging modalities help in the diagnosis of residual cholesteatoma. Diffusion weighted magnetic resonance imaging play an important role in diagnosis of retraction pockets .

Diffusion weighted magnetic resonance imaging is based on the principle of random microscopic motion (Brownian motion) of water molecules.This "diffusion" of water molecules differs in each biological tissue, For example water molecules in cholesteatoma are less mobile giving rise to a hyper-intense signal, while in other tissues as granulation tissues, water molecules are more mobile thus appear less intense on diffusion weighted magnetic resonance imaging sequence.

ELIGIBILITY:
Inclusion Criteria:

* • all patients presented with suspected primary cholesteatoma ,high risk retraction pockets ,Suspected recurrent or residual cholesteatoma after surgery .

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (e.g., pacemaker, metallic implant,cochlear implant Or claustrophobia).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presented with suspected cholesteatoma in assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Detection of Cholesteatoma Using Diffusion Magnetic Resonance Imaging | with in one year
  To detect the ability of Diffusion Magnetic Resonance Imaging in detection of cholesteatoma as compared by post operative data

CONTACTS AND LOCATIONS:
Overall Officials: amer ragab, resident, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander AE Jr, Caldemeyer KS, Rigby P. Clinical and surgical application of reformatted high-resolution CT of the temporal bone. Neuroimaging Clin N Am. 1998 Aug;8(3):631-50. PMID 9673317
- [Background] Nevoux J, Lenoir M, Roger G, Denoyelle F, Ducou Le Pointe H, Garabedian EN. Childhood cholesteatoma. Eur Ann Otorhinolaryngol Head Neck Dis. 2010 Sep;127(4):143-50. doi: 10.1016/j.anorl.2010.07.001. Epub 2010 Aug 11. PMID 20860924
- [Background] Thomassin JM, Braccini F. [Role of imaging and endoscopy in the follow up and management of cholesteatomas operated by closed technique]. Rev Laryngol Otol Rhinol (Bord). 1999;120(2):75-81. French. PMID 10444978
- [Background] Blaney SP, Tierney P, Oyarazabal M, Bowdler DA. CT scanning in "second look" combined approach tympanoplasty. Rev Laryngol Otol Rhinol (Bord). 2000;121(2):79-81. PMID 10997063
- [Background] Vanden Abeele D, Coen E, Parizel PM, Van de Heyning P. Can MRI replace a second look operation in cholesteatoma surgery? Acta Otolaryngol. 1999;119(5):555-61. doi: 10.1080/00016489950180784. PMID 10478595
- [Background] Kimitsuki T, Suda Y, Kawano H, Tono T, Komune S. Correlation between MRI findings and second-Look operation in cholesteatoma surgery. ORL J Otorhinolaryngol Relat Spec. 2001 Sep-Oct;63(5):291-3. doi: 10.1159/000055760. PMID 11528272
- [Background] Bergui M, Zhong J, Bradac GB, Sales S. Diffusion-weighted images of intracranial cyst-like lesions. Neuroradiology. 2001 Oct;43(10):824-9. doi: 10.1007/s002340100595. PMID 11688697
- [Background] Alzahrani M, Saliba I. Tympanic membrane retraction pocket staging: is it worthwhile? Eur Arch Otorhinolaryngol. 2014 Jun;271(6):1361-8. doi: 10.1007/s00405-013-2644-4. Epub 2013 Jul 27. PMID 23892691
- [Background] Bammer R. Basic principles of diffusion-weighted imaging. Eur J Radiol. 2003 Mar;45(3):169-84. doi: 10.1016/s0720-048x(02)00303-0. PMID 12595101
- [Background] De Foer B, Vercruysse JP, Bernaerts A, Maes J, Deckers F, Michiels J, Somers T, Pouillon M, Offeciers E, Casselman JW. The value of single-shot turbo spin-echo diffusion-weighted MR imaging in the detection of middle ear cholesteatoma. Neuroradiology. 2007 Oct;49(10):841-8. doi: 10.1007/s00234-007-0268-3. Epub 2007 Sep 3. PMID 17768611